CLINICAL TRIAL: NCT03292471
Title: Immediate and Cumulative Effects of rTMS on Brain Activation in Chronic Aphasia
Brief Title: Effects of rTMS on Brain Activation in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2566-P; I21RX002566-01A1 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-25 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Aphasia, Acquired
Keywords: Aphasia; Rehabilitation; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive 10 sessions of inhibitory rTMS to right hemisphere pars triangularis (RH PTr), either preceded by a 6 Hz priming rTMS stimulation sequence or not.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Inhibitory only (Experimental): Inhibitory 1Hz rTMS will be applied continuously for 1200 pulses (20 minutes) 5 days per week across 2 weeks (10 sessions total).
  Interventions: Device: Transcranial Magnetic Stimulation
- Excitatory primed (Experimental): The inhibitory sequence described above will be preceded for each session by priming stimulation which will consist of intermittent 6-Hz rTMS applied in 5 second trains with 25 second intervals between trains for a total 600 pulses (10 minutes).
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — rTMS is a non-invasive brain stimulation technique in which a focal, time-varying magnetic field is applied to a specific brain area to induce neuronal depolarization. rTMS can be used to selectively target a given brain region with a resolution as focal as 0.5 cm3 .Typically, administering a slow (1 Hz) sequence of magnetic pulses via rTMS temporarily reduces cortical excitability in the targeted brain region.
  Other Names: rTMS

SUMMARY:
This study will investigate the use of repetitive transcranial magnetic stimulation (rTMS), a non-invasive brain stimulation method, to improve word-finding abilities in Veterans and non-Veterans with chronic language problems following stroke (aphasia). Improving word-finding is important because word-finding difficulties are among the most common and debilitating consequences of aphasia. Although rTMS has shown promise as a treatment approach, not all individuals with aphasia show the same level of benefit. Specifically, this study will use functional magnetic resonance imaging (fMRI) to examine whether the likelihood of improved word-finding abilities following rTMS depends on pre-intervention language-related brain activity and will examine changes in brain activity in response to stimulation. A better understanding of how and for whom rTMS works will 1) help to identify the best candidates for rTMS treatment, 2) optimize rTMS treatment protocols to improve patient outcomes, and 3) improve the investigators' understanding of how the brain re-organizes language functions following stroke.

DETAILED DESCRIPTION:
Aphasia, an acquired communication disorder, is a common consequence of left-hemisphere stroke. Persisting, or chronic, aphasia negatively impacts not only interpersonal communication but participation in activities of daily living, independence, and autonomy. It is also associated with higher rates of depression and lower quality of life. Therefore, examining factors and treatments that result in the best possible recovery of language function for individuals with chronic aphasia is of paramount importance.

An intervention approach that has shown promise in early-phase research on treatment of chronic aphasia is repetitive transcranial magnetic stimulation (rTMS). rTMS is a non-invasive brain stimulation technique that can be used to focally modulate activity in targeted brain regions. Studies have shown that multiple sessions of 1Hz inhibitory rTMS applied to the right hemisphere Pars Triangularis (PTr) of people with chronic aphasia results in improved naming abilities. These improvements accrue over time, and may persist even after rTMS has ended. It has been proposed that rTMS induces this improvement by reducing the disruptive influence of compensatory activity in the right hemisphere PTr, allowing for recruitment of more efficient left hemisphere peri-lesional brain areas. However, existing neuroimaging evidence to support this hypothesis is insufficient.

The goal of the proposed study is to investigate the neurological mechanisms underlying the effect of rTMS on naming performance in chronic aphasia. This will extend existing knowledge regarding hemispheric contributions to language recovery following stroke and elucidate how rTMS-induced neuroplasticity can be co-opted to encourage optimal reorganization. The study will also investigate a potential source of individual response variability to rTMS, one which can inform both candidate selection and optimal stimulation parameters. Sixteen participants will be enrolled, yielding a significantly larger sample size than previous studies that have examined changes in functional brain activation in response to rTMS (n = 1, 2).

All participants will receive a sequence of 1200 pulses of 1 Hz rTMS to right hemisphere PTr across 10 daily sessions. Half of the participants will also receive a 6 Hz rTMS excitatory priming pulse sequence immediately prior to the 1 Hz sequence. This priming sequence ensures a consistent inhibitory response to the subsequent 1Hz rTMS and will permit an examination of state-dependent individual response variability.

To evaluate the effect of rTMS over time, participants will undergo functional magnetic resonance (fMRI) scans at four time points: prior to initiation of rTMS ("baseline"), immediately following the first rTMS session ("post-rTMS"), following the conclusion of the rTMS series ("post-treatment") and at a 2-month follow-up visit. During the scans, participants will be asked to name pictures, and both patterns of regional naming-related activation and effective connectivity (directional causal influence between activated brain regions) will be evaluated at each time point. In addition, naming performance will be measured via standardized assessments at baseline, post-treatment, and follow-up.

Changes in naming performance will be assessed over time, as a measure of rTMS effectiveness overall and between groups (priming sequence vs no priming sequence). In addition, changes in activation and effective connectivity will be correlated with naming improvement to assess the relative effectiveness of right hemisphere recruitment compared to left hemisphere peri-lesional recruitment. Overall increases in left hemisphere recruitment are hypothesized to result in greater improvements. However, the magnitude of left hemisphere recruitment due to rTMS is expected to depend on baseline levels of right hemisphere PTr activity.

Results from this study will significantly improve the investigator's understanding of the effects of rTMS on stroke recovery. The results will also inform future studies evaluating rTMS as an adjunct to behavioral speech-language intervention, augmenting therapeutic gains from traditional aphasia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aphasia due to unilateral left-hemisphere stroke
* Greater than 6 months post aphasia onset
* English as a first language
* No contraindications to MRI or TMS including:

  * pregnancy
  * presence of ferromagnetic substances in the head with the exception of dental fillings, stents or aneurysm clips documented to be MRI compatible
  * presence of any implanted devices including cardiac pacemaker, implanted cardiac defibrillator, insulin pump, cochlear implant, or drug infusion device
  * history of epilepsy; use of medications that are known to lower seizure threshold
  * severe claustrophobia

Exclusion Criteria:

* History for progressive neurological disease or premorbid language disorder
* Presence of severe motor speech disorder
* Drug or alcohol dependence, or significant mood or behavioral disorder that is not currently stable or medically managed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L. Gravier, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to group assignment, participants completed the Comprehensive Aphasia Test to determine aphasia severity, as groups were pseudorandomized on this basis (groups were balanced for average aphasia severity). In addition, participants completed an MRI screener and medical records were reviewed to screen for the presence of contraindications to MRI and/or rTMS.
Groups:
- Inhibitory Only: Inhibitory 1Hz rTMS was applied continuously for 1200 pulses (20 minutes) 5 days per week across 2 weeks (10 sessions total).
- Excitatory Primed: The inhibitory sequence (1Hz rTMS was applied continuously for 1200 pulses) was preceded for each session by priming stimulation which consisted of intermittent 6-Hz rTMS applied in 5 second trains with 25 second intervals between trains for a total 600 pulses (10 minutes).
Period: Overall Study
Arm/Group | Inhibitory Only | Excitatory Primed
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Excitatory Primed: The inhibitory sequence (1Hz rTMS was applied continuously for 1200 pulses) was preceded for each session by priming stimulation which will consist of intermittent 6-Hz rTMS applied in 5 second trains with 25 second intervals between trains for a total 600 pulses (10 minutes).
- Total: Total of all reporting groups
Arm/Group | Inhibitory Only | Excitatory Primed | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16
Aphasia Severity (Comprehensive Aphasia Severity Mean Modality T-Score) [Mean (Standard Deviation); unit: T-Score] — CAT mean modality T-Score (average of all language subscale T-scores of the Comprehensive Aphasia Test) is a measure of overall aphasia severity. A T-score of 50 reflects mean performance for the CAT normative sample of individuals with aphasia, with a standard deviation of 10 (higher scores reflect better performance/less severe aphasia).
  T-Score | 53.56 (5.25) | 53.86 (4.29) | 53.64 (4.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in Philadelphia Naming Test (PNT) Performance
Description: The Philadelphia Naming Test is a performance-based measure commonly used to assess naming (word production) ability among adults with aphasia. The minimum raw score is 0 and the maximum is 175 (higher scores reflect more accurate naming/better naming ability).
Time Frame: Pre- to post treatment (an average of 3 weeks), and at 2 month follow-up
Population: 5 participants in each group were able to return for 2-month follow up testing
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Inhibitory Only | Excitatory Primed
Number analyzed (Participants) | 8 | 8
Score on a scale
  Pre-treatment | 122.125 (27.18) | 130.875 (22.86)
  Post-treatment | 132.5 (28.65) | 142.125 (16.71)
  Follow-up: number analyzed (Participants) | 5 | 5
  Follow-up | 115.6 (21.85) | 133.6 (26.84)
Statistical Analysis 1: Comparison: Inhibitory Only vs Excitatory Primed; Baysian Multivariate Analysis of Variance; Test type: Superiority — Dependent variable: PNT T-score Fixed Effects: Group Assignment (A = Standard, B= Priming), Time point (Pre-treatment, Post-treatment) Random Effects: Participant (intercept and slope) Priors for slope and intercept were set as t-distributions (PNT raw score converted to T-score scale with m = 50, sd = 10 based on sample estimates from Fergadiotis, Hula, & Kellough, 2015); Highest Density Interval of Posterior Di = .284, 95% CI 2-sided [-2.07 to 2.92] — Direction of comparison: Group A (Standard Protocol) and post-treatment timepoint were set as reference values
Statistical Analysis 2: Comparison: Inhibitory Only vs Excitatory Primed; Baysian Multivariate Analysis of Variance; Test type: Superiority — Dependent variable: PNT T-score Fixed Effects: Group Assignment (A = Standard, B= Priming), Time point (Pre-treatment, Follow-up) Random Effects: Participant (intercept and slope) Priors for slope and intercept were set as t-distributions (PNT raw score converted to T-score scale with m = 50, sd = 10 based on sample estimates from Fergadiotis, Hula, & Kellough, 2015); Highest Density Interval of Posterior Di = .02, 95% CI 2-sided [-2.38 to 2.46] — Direction of comparison: Group A (Standard Protocol) and follow-up (2 months post-treatment) timepoint were set as reference values

2. Secondary Outcome: Change in Comprehensive Aphasia Test (CAT) Performance
Description: The Comprehensive Aphasia Test is a performance-based measure of language processing across multiple language domains commonly used to assess language-processing ability among adults with aphasia. CAT mean modality T-Score (average of all language subscale T-scores of the Comprehensive Aphasia Test) is a measure of overall aphasia severity. A T-score of 50 reflects mean performance for the CAT normative sample of individuals with aphasia, with a standard deviation of 10 (higher scores reflect better performance/less severe aphasia).
Time Frame: Pre- to post treatment (an average of 3 weeks), and at 2 month follow-up
Population: 5 participants in each group were able to return for follow-up testing
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Inhibitory Only | Excitatory Primed
Number analyzed (Participants) | 8 | 8
T-Score
  Pre-treatment | 53.56 (5.25) | 53.875 (4.29)
  Post-treatment | 54.54 (5.45) | 55.71 (4.59)
  Follow-up: number analyzed (Participants) | 5 | 5
  Follow-up | 52.5 (4.04) | 56.7 (5.3)
Statistical Analysis 1: Comparison: Inhibitory Only vs Excitatory Primed; Baysian Multivariate Analysis of Variance; Test type: Superiority — Dependent variable: CAT Mean-modality T-score Fixed Effects: Group Assignment (A = Standard, B= Priming), Time point (Entry, Exit) Random Effects: Participant (intercept and slope) Priors for slope and intercept were set as t-distributions; Highest Density Interval of Posterior Di = .997, 95% CI 2-sided [-0.0719 to 2.25] — Direction of comparison: Group A (Standard Protocol) and post-treatment timepoint were set as reference values
Statistical Analysis 2: Comparison: Inhibitory Only vs Excitatory Primed; Baysian Multivariate Analysis of Variance; Test type: Superiority — Dependent variable: CAT Mean-modality T-score Fixed Effects: Group Assignment (A = Standard, B= Priming), Time-point (Pre-treatment, Post-treatment) Random Effects: Participant (intercept and slope) Priors for slope and intercept were set as t-distributions; Highest Density Interval of Posterior Di = .443, 95% CI 2-sided [-0.596 to 1.58] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Approximately 3 months
Description: An adverse event reporting form was completed at each assessment and treatment visit
Arm/Group | Inhibitory Only | Excitatory Primed
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhibitory Only (N=8) | Excitatory Primed (N=8)
Mild Headache (General disorders) | 0 | 1 (3)

LIMITATIONS AND CAVEATS:
Unable to collect all planned functional MRI data due to technical difficulties/scanner out of service.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03292471/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT03292471/ICF_001.pdf